CLINICAL TRIAL: NCT00359593
Title: Stroke Canada Optimization of Rehabilitation by Evidence Implementation Trial (SCORE IT)
Brief Title: Stroke Canada Optimization of Rehabilitation by Evidence Implementation Trial SCORE-IT)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CSNscore
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2006-07

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Knowledge translation; Evidence based practice; Outcomes
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Behavioral: Knowledge translation intervention package

SUMMARY:
The aim of this project is to evaluate whether using an implementation intervention promotes use of best practices by rehabilitation professionals and leads to improvements in patient outcomes for individuals with stroke.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability in Canada and frequently causes hemiparesis (upper limb and lower limb weakness on one side of the body). Approximately one third of stroke survivors require physical rehabilitation to improve their motor and functional recovery (1). Although many strategies have been shown to be effective in promoting recovery after stroke, the uptake of evidence-based practice by rehabilitation professionals across Canada is variable. The aim of this project is to evaluate whether using an implementation intervention promotes use of best practices by rehabilitation professionals and leads to improvements in patient outcomes for individuals with stroke.

This project is a cluster randomized implementation trial for upper and lower limb interventions. Rehabilitation centres across Canada will be randomized to receive either an outcome-oriented implementation strategy (OOI) to facilitate implementation of the EIPRs or a process-oriented implementation strategy (POI). At the onset, rehabilitation professionals practicing in all centres will receive education in using best practice outcome measures related to stroke rehabilitation. All centres will be assessed for baseline adherence to the EIPRs. Centres in the OOI will receive "usual care" (i.e. passive dissemination of the written protocols and information about outcome measures). Centres in the POI arm will receive a combination of strategies to facilitate EIPR uptake (i.e., use of a local facilitator, practice audits with feedback, reminder systems and educational sessions). Following exposure to the EIPRs, all centres will document adherence to the EIPRs, and patient outcomes as assessed by the measures. An analysis of the costs associated with rehabilitation interventions and the incremental expense of a POI strategy will be undertaken. These data will be used to compare the OOI and POI centres with respect to the level of uptake and implementation of EIPRs and related expenses.

ELIGIBILITY:
Rehabilitation Hospitals/Research Sites:

Inclusion Criteria:

* hospital with designated rehabilitation beds;
* regularly treats stroke patients;
* has access to at least one physical (PT) and one occupational (OT) therapist on the health professional team

Exclusion Criteria:

* Inadequate staffing to administer the outcome measures consistently

Patients:

Inclusion Criteria:

* medically stable;
* stroke with residual disability;
* requires complex rehabilitation interventions from at least 3 health care professionals, one of them being an OT or a PT;
* admitted to rehabilitation centre within 90 days of stroke onset;
* and age >18 years

Exclusion Criteria:

* having a medical condition that is expected to result in death within 6 months;
* presence of a serious chronic disabling condition that impacts on either the rehabilitation process or rehabilitation outcomes such as severe arthritis, dementia, Parkinson's disease;
* active suicidal ideation or symptoms of psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2006-09; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Arm function as measured by the Box and Block test
Walking speed as measured by the 6 minutes walk test

SECONDARY OUTCOMES:
Arm function as measured by the Chedoke Arm and Hand Activity Inventory (CAHAI- 9)
Impairment as measured by the Chedoke-McMaster Stroke Assessment Scale (CMSA)
Independence of daily living as measured by the 3. Functional Independence Measure (FIM)
Economic outcomes measured by the Quality Adjusted Life Years (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Bayley, MD, Principal Investigator — Toronto Rehabilitation Institute; Sharon Wood-Dauphinee, PhD, Principal Investigator — McGill University
Locations (2):
- Canada (2):
  - Toronto Rehabilitation Institute, Toronto, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Salbach NM, Wood-Dauphinee S, Desrosiers J, Eng JJ, Graham ID, Jaglal SB, Korner-Bitensky N, MacKay-Lyons M, Mayo NE, Richards CL, Teasell RW, Zwarenstein M, Bayley MT; Stroke Canada Optimization of Rehabilitation By Evidence - Implementation Trial (SCORE-IT) Team. Facilitated interprofessional implementation of a physical rehabilitation guideline for stroke in inpatient settings: process evaluation of a cluster randomized trial. Implement Sci. 2017 Aug 1;12(1):100. doi: 10.1186/s13012-017-0631-7. PMID 28764752
- See also: Canadian Stroke Network — http://www.canadianstrokenetwork.ca/eng/index_flash.php